CLINICAL TRIAL: NCT01844674
Title: A Phase I, Open-Label, Multicenter, 3- Period, Fixed-Sequence Study to Investigate the Effect of Vemurafenib on the Pharmacokinetics of a Single Dose of Tizanidine (a CYP1A2 Substrate) in Patients With BRAFV600 Mutation-Positive Metastatic Malignancy
Brief Title: A Study on the Effect of Vemurafenib on the Pharmacokinetics of a Single Dose of Tizanidine in Patients With BRAFV600 Mutation-Positive Metastatic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GO28396; 2012-003705-94 (EudraCT Number)
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Malignant Melanoma, Neoplasms
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — tizanidine; Vemurafenib

ARMS (1):
- Pharmacokinetic Population (Experimental): All participants will receive a 3-period treatment including single-dose tizanidine on Day 1, twice-daily vemurafenib on Days 2 to 21, and both agents together on Day 22.
  Interventions: Drug: Tizanidine; Drug: Vemurafenib

INTERVENTIONS:
Drug: Tizanidine — Participants will receive tizanidine as single oral doses, 2 milligrams (mg) on Day 1 and repeated on Day 22, each following an overnight fast >/= 10 hours.
Drug: Vemurafenib — Participants will receive vemurafenib as multiple oral doses, 960 mg twice daily on Days 2 to 22.

SUMMARY:
This open-label, multicenter, 3-period, fixed-sequence study will evaluate the effect of multiple oral doses of vemurafenib on the pharmacokinetics of a single oral dose of tizanidine in participants with BRAFV600 mutation-positive metastatic malignancies. Participants will receive a single oral dose of tizanidine on Day 1, vemurafenib orally twice daily on Days 2 to 21, and tizanidine and vemurafenib on Day 22. Eligible participants will have the option to continue treatment with vemurafenib as part of an extension study (NCT01739764).

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 70 years of age, inclusive
* Unresectable Stage IIIc or IV metastatic melanoma positive for the BRAFV600 mutation or other malignant tumor type which harbors a V600 activating mutation of BRAF, as determined by Cobas 4800 BRAFV600 Mutation Test or a DNA sequencing method
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Life expectancy greater than or equal to (>/=) 12 weeks
* Participant has not consumed tobacco or nicotine-containing products for 42 days prior to first dose of study drug, and must agree to refrain from such products while on study
* Adequate hematologic, renal and liver function

Exclusion Criteria:

* Prior treatment with vemurafenib or other BRAF inhibitor within 42 days of Day 1
* History of or current clinically significant cardiac or pulmonary dysfunction, including current uncontrolled Grade >/= 2 hypertension or unstable angina
* Current dyspnea at rest due to complications of advanced malignancy or any requirement for supplemental oxygen
* Active central nervous system lesions (participants with radiographically unstable, symptomatic lesions)
* Participants with CYP1A2 gene mutation (-3113G->A), either in one or two alleles
* Allergy or hypersensitivity to vemurafenib or tizanidine formulations
* Current severe uncontrolled systemic disease
* Inability or unwillingness to swallow pills
* History of malabsorption or other condition that would interfere with enteral absorption of study treatment
* History of clinically significant liver disease (including cirrhosis), current alcohol abuse, or human immunodeficiency (HIV) infection requiring antiretroviral treatment, acquired immune deficiency syndrome (AIDS)-related illness, or active hepatitis B or C
* Pregnant or breastfeeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09-02 (Actual); Primary Completion 2014-08-26 (Actual); Study Completion 2014-08-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of tizanidine under conditions of vemurafenib steady-state exposure: Area under the concentration-time curve (AUC) | Pre-dose and up to 12 hours post-dose
Pharmacokinetics of tizanidine under conditions of vemurafenib steady-state exposure: Maximum plasma concentration (Cmax) | Pre-dose and up to 12 hours post-dose
Pharmacokinetics of tizanidine under conditions of vemurafenib steady-state exposure: Time to maximum plasma concentration (Tmax) | Pre-dose and up to 12 hours post-dose
Pharmacokinetics of tizanidine under conditions of vemurafenib steady-state exposure: Terminal half-life (t1/2) | Pre-dose and up to 12 hours post-dose
Pharmacokinetics of tizanidine under conditions of vemurafenib steady-state exposure: Apparent clearance (CL/F) | Pre-dose and up to 12 hours post-dose

SECONDARY OUTCOMES:
Safety: Incidence, nature and severity of adverse events and serious adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 | Up to approximately 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (3):
  - Diablo Valley Oncology and Hematology, Pleasant Hill, California
  - Karmanos Cancer Center, Detroit, Michigan
  - Duke University Health Systems, Durham, North Carolina
- Brazil (4):
  - Instituto Nacional do Cancer - INCA, Rio de Janeiro, Rio de Janeiro
  - Hospital de Caridade de Ijui; Oncologia, Ijuí, Rio Grande do Sul
  - CITO - Centro Integrado de Terapia Onco-Hematológica - Hospital da Cidade de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
- CSSS champlain - Charles-Le Moyne, Greenfield Park, Quebec, Canada
- Bank of Cyprus Oncology Center, Nicosia, Cyprus
- South Korea (3):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center., Seoul